CLINICAL TRIAL: NCT01358903
Title: Open-Label Multicenter 2-Arm Phase I Study of RO5429083 With Dose-Escalation and Extension Cohorts, and Imaging Cohorts With RO5429083 and 89Zr-labeled RO5429083, in Patients With Metastatic and/or Locally Advanced, CD44-Expressing, Malignant Solid Tumors
Brief Title: A Study of RO5429083 in Patients With Metastatic and/or Locally Advanced, CD44-Expressing, Malignant Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP25385; 2010-021168-13 (EudraCT Number)
Record Dates: First submitted 2011-05-18; First posted 2011-05-24 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

ARMS (2):
- A (Experimental)
  Interventions: Drug: RO5429083
- B (Experimental)
  Interventions: Drug: RO5429083

INTERVENTIONS:
Drug: RO5429083 — Cohorts receiving multiple escalating doses iv
  Arms: A
Drug: RO5429083 — Cohorts receiving 89Zr-labelled RO5429083 plus RO5429083, followed by RO5429083 until disease progression
  Arms: B

SUMMARY:
This open-label 2-arm study will assess the pharmacokinetics, pharmacodynamics, safety and efficacy of RO5429083 in patients with metastatic and/or locally advanced CD44-expressing malignant solid tumors. In Part A, cohorts of patients will receive RO5429083 intravenously at escalating doses. In Part B, patients will receive 89Zr-labelled RO5429083 in Cycles 1 and/or 2, followed by RO5429083. For all patients there will be an option to continue treatment with RO5429083 until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Metastatic and/or locally advanced malignant CD44-expressing solid tumors
* Patients with disease progression on standard therapy, or have tumors that are not curable by standard therapy
* Life expectancy of over 12 weeks

Exclusion Criteria:

* Concurrent therapy with any other investigational drug
* Known or suspected CNS metastases including leptomeningeal metastases
* Active bleeding, bleeding diathesis or history of coagulation disorder
* Uncontrolled diabetes mellitus
* Active or uncontrolled infections
* Patients with HIV infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2011-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Arm A: Safety (Incidence of adverse events related to study drug) | Until disease progression or unacceptable toxicity (approximately 2 years)
Arm A: Maximum tolerated dose of RO5429083 | Until disease progression or unacceptable toxicity (approximately 2 years)
Arm A: Tumor Growth Control Rate | Until disease progression or unacceptable toxicity (approximately 2 years)
Arm B: Tissue distribution of RO5429083 assessed by positron emission tomography (PET) | Until disease progression or unacceptable toxicity (approximately 2 years)
Arm A: Pharmacokinetics (serum levels of RO5429083) | Until disease progression or unacceptable toxicity (approximately 2 years)

SECONDARY OUTCOMES:
Arm A: Recommended dose of RO5429083 for the extension cohort | Until disease progression or unacceptable toxicity (approximately 2 years)
Arm A: Anti-tumor activity of RO5429083 | Until disease progression or unacceptable toxicity (approximately 2 years)
Arm B: Target saturation of 89Zr-labelled RO5429083 | Until disease progression or unacceptable toxicity (approximately 2 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- United States (2):
  - Houston, Texas
  - Seattle, Washington
- France (2):
  - Paris
  - Toulouse
- Netherlands (2):
  - Amsterdam
  - Nijmegen